CLINICAL TRIAL: NCT06563947
Title: A Clinical Study to Evaluate the Effectiveness of Oral Enterobacterial Capsules in Patients With Intermediate and Advanced HCC Who Have Progressed After Immune Checkpoint Inhibitor Combination With Anti-Angiogenesis Targeted Agents
Brief Title: Single Arm Clinical Trial (Gut Microbiota and HCC)
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xu Yong, MD (Other)
Collaborators: Nanjing Xiershou Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor-Investigator, Xu Yong, MD, Secretary of the Party Committee & Principal Investigator, Shenzhen Third People's Hospital
Organization: Shenzhen Third People's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY2024-178
Record Dates: First submitted 2024-08-14; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-center, single-arm clinical study. For those who meet the enrollment conditions, the original regimen of immune checkpoint inhibitors combined with anti-angiogenic targeted drugs will remain unchanged after enrollment.On this basis, the study subjects started oral enterobacterial capsules to see whther enterobacterial capsules could improve the efficacy of patients receiving the above treatment regimens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with progressed HCC after treatment were given enterobacterium capsules (Experimental): Patients were given oral enterobacterium capsules (300 mg/per capsule) 6 capsules/day for 10 consecutive days, and then discontinued to the next course of treatment.
  Interventions: Biological: Oral enterobacterium capsules

INTERVENTIONS:
Biological: Oral enterobacterium capsules — Enterobacterium capsules (300 mg/per capsule) orally 6 capsules/day for 10 consecutive days.

SUMMARY:
To evaluate the efficacy and safety of oral enterobacterial capsules in patients with intermediate and advanced HCC who have progressed after treating with immune checkpoint inhibitors in combination with anti-angiogenesis targeted agents.

DETAILED DESCRIPTION:
This is a prospective, single-center, single-arm clinical study. For those who meet the enrollment conditions, the original regimen of immune checkpoint inhibitors combined with anti-angiogenic targeted drugs will remain unchanged after enrollment.On this basis, the study subjects started oral enterobacterial capsules to see whther enterobacterial capsules could improve the efficacy of patients receiving the above treatment regimens.

Oral administration of intestinal bacteria capsules 6 capsules/day, after observing no adverse reactions, oral administration for 10 consecutive days, 6 capsules/day from the second day to the tenth day, and then discontinued to the next course of treatment.

Total course of treatment: a total of 4 courses of oral intestinal bacteria capsules, each course of oral administration for 10 days, and a course of 21 days; A course of TKI combined with immune checkpoint inhibitors treatment is 21 days until the disease progresses or intolerable toxicity and side effects appear.

Observe the metrics: Primary Clinical Endpoint - Progression-Free Survival (PFS); Secondary Clinical Endpoints - Overall Growth Phase (OS), Objective Response Rate (ORR), Duration of Response (DOR), and Disease Control Rate (DCR). The new RECIST1.1 criteria were used for the efficacy evaluation system, the CTCAE5.0 grading system was used for the evaluation of common adverse reactions during treatment, and other indicators included imaging including conventional biochemical indexes such as CT and ultrasound, as well as quality of life scores.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, gender is not limited;
2. Confirmed imaging or histological diagnosis of unresectable HCC, BCLC stadium B or C;
3. Clinical diagnosis of HCC progression during TKIs combined with ICIs treatment;
4. Not suitable for local ablation or chemoembolization;
5. Child-Pugh Grade A;
6. ≥ 1 measurable lesion (RECIST v1.1)
7. ECOG PS 0-1

Exclusion Criteria:

1. Usage of antibiotics within 2 weeks prior enrollment;
2. Diagnosis of immunodeficiency (e.g. HIV, immunosuppressants)
3. Patients with known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation;
4. Female patients who are pregnant or breastfeeding;
5. Patients with untreated acute or chronic active hepatitis B or hepatitis C infection.
6. Patients are currently undergoing clinical trials of other drugs;
7. Patients are considered by the investigator to be unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-08-24 (Estimated); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Objective Progression-Free Survival (PFS) | Up to approximately 1 years
  To analyse the Progression-Free Survival (PFS) of patients
Objective Secondary Clinical Endpoints - Overall Growth Phase (OS) | Up to approximately 1 years
  To analyse the Secondary Clinical Endpoints - Overall Growth Phase (OS) of patients
Objective Objective Response Rate (ORR) | Up to approximately 1 years
  To exprole the Objective Response Rate (ORR) of patients
ObjectiveDuration of Response (DOR) | Up to approximately 1 years
  To analyse the Duration of Response (DOR) of patients
Diversity analysis | Up to approximately 1 years
  We will use 16S rRNA sequencing to measure fecal sample. The alpha and beta diversity of gut microbiota will be analyzed, including a series of statistical analysis indexes such as Chao, Shannon, Simpsonace, Simpson and Coverage, in order to reflect the microbial community diversity.
Species differential analysis | Up to approximately 1 years
  We will use 16S rRNA sequencing to measure fecal sample. Based on the results of species annotation, the PCA、PCoA and NMDS analysis will be used to assess the similarities and differences in species composition.
Feces Metabolomics | Up to approximately 1 years
  Changes of metabolites in feces measured by metabolomic mass spectrometry, unsupervised PCA (principal component analysis) was performed by statistics function prcomp, identified metabolites were annotated using KEGG Compound database.
Serum Metabolomics | Up to approximately 1 years
  Changes of metabolites in serum measured by metabolomic mass spectrometry, unsupervised PCA (principal component analysis) was performed by statistics function prcomp, identified metabolites were annotated using KEGG Compound database.

CONTACTS AND LOCATIONS:
Overall Officials: Yong Xu, Dr, Principal Investigator — Secretary of the Party Committee of the Shenzhen Third People's Hospital

IPD SHARING:
Plan to Share IPD: No